CLINICAL TRIAL: NCT05825352
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "Ocular Drops Based Upon Carmellose" Used to Relieve Dry Eye Symptoms
Brief Title: PMCF Study to Evaluate Performance and Safety of "Ocular Drops Based Upon Carmellose" Used to Relieve Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R4-CMC
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye; Dry Eye Disease; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Carmellose eye drops

INTERVENTIONS:
Device: Carmellose eye drops — Ocular drops based upon carmellose

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a multifactorial disease of the ocular surface characterized by loss of homeostasis of the tear film and accompanied by symptoms such as ocular discomfort and visual disturbance.

Tear Film & Ocular Surface Society Dry Eye Workshop (TFOS DEWS) II recommends individualized management of DED based on the relative contribution of aqueous deficient and evaporative pathophysiology (to the extent that this can be determined), as well as disease severity.

First-line for treating dry eye consists of over the counter (OTC) artificial tear drops, gels, ointments, or lubricants.

Carboxymethyl cellulose (CMC) is one of the most common viscous polymers used in artificial tears to achieve prolonged residence time on the ocular surface.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Ocular drops based upon carmellose" used as intended to relieve dry eye symptoms.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "Ocular drops based upon carmellose" according the Instructions for Use (IFU).

Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), one of the "Ocular drops based upon carmellose" products can be dispensed to the enrolled subject, depending on Investigator clinical evaluation and decision.

The patient will perform 2 on site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

The first administration and the intervals at which the treatment should be repeated, to be done as per Investigator judgment and according the IFU, depend on various factors regarding the physiology of the patients (e.g. type of eye-tear film, anatomy, age), their lifestyle (e.g. use of computer, wearing of contact lenses) and their eye-surgery history (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* Male and Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with ocular symptoms such as burning, itching, and foreign body sensation due to environmental factors, contact lenses wearing and/or mild-severe dry eye;
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Known hypersensitivity or allergy to Investigational Product (IP) components;
* Suspected alcohol or drug abuse;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I: to evaluate the lubricant and protecting performance of the "Ocular drops based upon carmellose" used as Intended in subjects with mild or severe dry eye syndrome, through the Schirmer I test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)

SECONDARY OUTCOMES:
Change in Tear Break-up Time (TBUT): to evaluate the performance of the "Ocular drops based upon carmellose" used as Intended to ensure relief from ophthalmic stress, through the TBUT test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
Change in Ocular Surface Disease Index (OSDI): to evaluate the eye-discomfort relieving performance of the "Ocular drops based upon carmellose", through OSDI | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
To evaluate the safety and tolerability of the "Ocular drops based upon carmellose", through Visual Analogue Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness) | End of study visit (EOS/V2 = Day 30 ± 2)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the patient satisfaction through a Rensis Likert 5 points patient satisfaction scale | End of study visit (EOS/V2 = Day 30 ± 2)
  Rensis Likert 5 points patient satisfaction scale:
  Minimum value: Very dissatisfied Maximum value: Very satisfied High score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy